CLINICAL TRIAL: NCT06780033
Title: A Phase 1, Randomized, Double-blind, Placebo Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ART101 in Adult Participants With Hypertension.
Brief Title: A Study to Evaluate ART101 in Adult Participants With Hypertension
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: At Sponsor's Request
Sponsor: Arnatar Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ART101-C101
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ART101 SAD (Experimental): Participants will receive single subcutaneously of ART101 or placebo on day 1 following a minimum of 8-hour fast.
  Interventions: Drug: ART-101 - SAD
- Placebo (Placebo Comparator): Participants will receive a single dose subcutaneously of placebo on day 1 following a minimum of 8-hour fast.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ART-101 - SAD — Forty participants will be enrolled across 5 SAD cohorts. The planned doses across 5 cohorts are as follows- include 20mg (SAD Cohort 1), 60mg (SAD Cohort 2). 150mg (SAD Cohort 3). 300mg (SAD Cohort 4) and 500 mg (SAD Cohort 5).
  Arms: ART101 SAD
Other: Placebo — Participants will receive matching placebo subcutaneously on Day 1 after 8 hour fast.
  Arms: Placebo

SUMMARY:
This is a Phase 1, first-in-human, randomized, double-blind, placebo-controlled, study to assess the safety, tolerability, Pharmacokinetics (PK), and pharmacodynamics (PD) of a single dose of ART101 administered via subcutaneous injection to hypertensive adult participants. An anticipated 5 dose cohorts (one as optional) with maximum of 40 participants will be randomized in SAD study.

DETAILED DESCRIPTION:
The study will be conducted across 5 single ascending dose (SAD) cohorts with approximately 40 participants.

Estimated study duration for each participant: Approximately 13.5 months including a 1.5-month Screening Period, 3-month Treatment Period and up to 12-month Follow-up post dose. On Day 1, participants will receive study drug as a single subcutaneous injection following a minimum 8-hour fast. The planned ART101 dose across 5 cohorts are as follows- 20mg, 60mg, 150mg, 300mg and 500mg. An SRC meeting will be held prior to dose escalations or prior to initiation of next cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (excluding women of child bearing potential [WOCBP]) aged 18 to 65 years (inclusive at the time of informed consent).
2. Hypertensive but otherwise in good general health, with no clinically significant medical history, and have no clinically significant abnormalities on physical examination at Screening and/or before the first administration of study drug at the discretion of the PI.
3. Either of the following:

   1. Drug Naïve.
   2. Has previously received monotherapy or dual therapy for hypertension but has ceased medication(s) under the supervision of the participant's medical professional eg, General Practitioner or Specialist.

   Note: Where applicable, a participant must have ceased administering therapy for hypertension from ≥ 3 weeks prior to Screening.
4. Mean sitting SBP > 130 mmHg and ≤ 159 mmHg per USA guidelines at Screening (by oscillometric AOBP measurement).

   Note: If the PI (or designee) considers that the Screening oscillometric AOBP measurement is spuriously elevated, oscillometric AOBP may be retested once during Screening.
5. Mean SBP > 130 mmHg and ≤ 159 mmHg from the daytime BP measurements and a night-time mean SBP ≥ 110mg Hg at Baseline per USA guidelines (assessed by 24-hour ABPM during the Screening Period) without hypertensive medication.

   Note: Where the PI (or designee) is informed that the 24-hour ABPM has failed quality check, the 24-hour ABPM may be repeated once during the Screening Period.
6. BMI between ≥ 18.0 and ≤ 35.0 kg/m2 at Screening and weight ≥ 50 kg at Screening.
7. Nonsmoker and must not have used any nicotine-containing products within 6 months prior to Screening.
8. ECG findings at Screening within normal range, unless deemed not clinically significant by the PI or designee.
9. Males must be surgically sterile vasectomized since at least 6 months prior to first study drug administration, OR if not surgically sterile AND will engage in sexual relations with a WOCBP, his female partner must meet 1 of the following criteria:

   1. Surgically sterile (eg, bilateral tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy, bilateral tubal ligation) or postmenopausal.
   2. Agree to use acceptable, highly effective, double barrier contraception from Screening until study completion, including the Follow-up Period. Acceptable, highly effective, double barrier contraception is defined as meeting 1 of the following criteria:

   i. Simultaneous use of hormonal contraceptives (implant, injection, pills, vaginal rings and skin patches) and must agree to use the same hormonal contraceptive throughout the study, and condom for the male participant.

   ii. Simultaneous use of Intrauterine Device (IUD) or Intrauterine System (IUS) (Mirena or Kyleena) and condom for the male participant.

   iii. Simultaneous use of diaphragm or cervical cap and male condom for the male participant.

   Note: Males with same-sex partners (abstinence from penile-vaginal intercourse) or are abstinent from heterosexual intercourse are not required to use contraception when this is their preferred and usual lifestyle. Note: Males must be willing not to donate sperm from the first dose of study drug until at least 90 days after study completion.
10. Able and willing to comply with study procedures, study restrictions, and visits to the study site.
11. Able and willing to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.

Exclusion Criteria:

1. WOCBP or female who is pregnant, breastfeeding, or planning to become pregnant during the study.
2. Mean sitting DBP > 110 mmHg at Screening (by oscillometric AOBP measurement) without hypertensive medication.
3. History of secondary hypertension including, but not limited to, any of the following:

   1. Renovascular hypertension (unilateral or bilateral renal artery stenosis).
   2. Coarctation of the aorta.
   3. Primary hyperaldosteronism.
   4. Cushing's disease, pheochromocytoma.
   5. Polycystic kidney disease.
   6. Drug induced hypertension.
4. Any of the following:

   1. Postural tachycardia (ie, > 30 bpm upon standing).
   2. Orthostatic hypotension (ie, a fall in SBP of ≥ 20 mmHg or DBP of ≥ 10 mmHg within 1 minute of standing up from a supine position).
   3. History of hypotension.
   4. Arm circumference does not align with any blood pressure cuff size. Note: Where applicable, a participant must have ceased administering monotherapy or dual therapy for hypertension from ≥ 3 weeks prior to Screening.

   Note: The relevant Australian Product Information should be reviewed by the PI or designee to determine the appropriate washout period for a prescription medication.

   Note: Cessation of prescription medication (eg, monotherapy or dual therapy for hypertension) by participant must occur with the approval of the participant's medical professional eg, General Practitioner or Specialist.
5. Diagnosed with diabetes mellitus.
6. Is participating in a concurrent experimental therapy study with a study drug or medical device.
7. Any of the following:

   1. Has received experimental therapy with a small molecule within 30 days of the first administration of study drug or 5 half-lives of the small molecule experimental therapy (whichever is the longer). Note: Experimental therapy with a small molecule refers to any small molecule compound (eg, Lipitor, Benadryl) under investigation in a clinical trial.
   2. Has received experimental therapy with a large molecule within 90 days of the first administration of study drug or 5 half-lives of the large molecule experimental therapy (whichever is the longer).

      Note: Experimental therapy with a large molecule refers to a large molecule (eg, monoclonal antibodies, peptides) under investigation in a clinical trial.
   3. Has received experimental therapy with antisense oligonucleotides or siRNA within 12 months of the first administration of study drug or 5 half-lives (whichever is longer).
   4. Has participated in more than 4 experimental therapy studies with an experimental therapy or medical device within 1 year prior to first administration of study drug.
   5. Has received any immune suppressing drug (including experimental therapies as part of a clinical study) within 4 months of the first administration of study drug or 5half-lives, whichever is longer.
8. Evidence or history of any clinically significant immunologic, hematologic, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, musculoskeletal, hepatic, psychiatric, neurologic, allergic disease (including clinically significant or multiple drug allergies), surgical conditions, or any condition that, in the opinion of the PI, that would jeopardize the safety of the participant, prevent complete participation in the study, or compromise interpretation of study data.
9. History of allergic reaction to an oligonucleotide, GalNAc-containing medication, or the study drug or its constituents.
10. History or presence of a condition associated with significant immunosuppression.
11. History of life-threatening infection (eg, meningitis).
12. History of malignancy, except for the following:

    1. Basal or squamous cell carcinoma of the skin excised more than 2 years prior to Screening.
    2. Cancer that has been resolved or has been in remission for more than 5 years prior to Screening.
13. History of porphyria, myopathy, cardiac valve repair, cardiac device implantation or an active liver disease (including steatotic hepatitis and fibrosis).
14. Has undergone surgical procedures within 4 weeks of Day -1, or is planning elective surgery until the angiotensinogen level has returned to >50% predose Baseline level or until at least Day 365 whichever comes first.
15. Unstable / underlying cardiovascular disease defined as:

    1. Any history of congestive heart failure (New York Heart Association [NYHA] Class III-IV).
    2. Any history of previous myocardial infarction, coronary revascularization, unstable or stable angina pectoris ˂ 6 months prior to Screening.
    3. Any hemodynamically unstable atrial or ventricular arrhythmias.
    4. Significant uncorrected valvular heart disease.
    5. History of stroke or transient ischemic attack < 6 months prior to Screening.
16. A cardiac valve repair, cardiac device implantation, and/or a hospitalization for heart failure within 3 months of Screening.
17. Any of the following:

    1. A personal or family history of long QT syndrome, Torsades de Pointes, or other complex ventricular arrhythmias, or family history of sudden death.
    2. History of, or current, clinically significant arrhythmias as judged by the PI, including ventricular tachycardia, ventricular fibrillation, atrial fibrillation, sinus node dysfunction, or clinically significant heart block. Participants with minor forms of ectopy (eg, premature atrial contractions) are not necessarily excluded.
    3. Abnormal ECG findings at Screening that are considered by the PI or designee to be clinically significant.
18. Any of the following:

    1. Evidence of severe acute respiratory syndrome-related coronavirus-2 (SARS-CoV-2) infection at Screening. During the study, a participant with an infection may continue the study at the discretion of the PI.
    2. Oral temperature > 38 °C on Day-1.
    3. Has experienced fever (body temperature > 38°C) or symptomatic viral or bacterial infection within 2 weeks prior to Screening.
    4. Has experienced any illness within 4 weeks of Day -1 deemed by the PI to be clinically significant.

    Has experienced infection within 3 months prior to Screening that required parenteral antibiotics.
19. Vaccination with a live vaccine (eg, MMR, rotavirus) within 4 weeks prior to the first administration of study drug.

    Note: Other exclusions pertaining to vaccination will be per PI discretion, in consultation with the Sponsor.
20. Aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma-glutamyl transferase, and/or bilirubin (total, direct, indirect) values > 1.5 × upper limit of normal at Screening. Bilirubin levels above > 1.5 x upper limit of normal will be acceptable, if they are consistent with Gilbert's syndrome, according to PI discretion. Repeat testing at Screening is acceptable for out-of-range values following approval by the PI or designee.
21. Positive test for HIV antibody, hepatitis C virus antibody, hepatitis B surface antigen.
22. Any clinically significant laboratory values (based on laboratory normal range) in the opinion of the Investigator. Repeat testing at Screening is acceptable for out-of-range values following approval by the PI or designee.
23. Estimated glomerular filtration rate (eGFR) of < 60 mL/min/1.73m2 (using the MDRD formula).
24. Blood donation > 500 mL, significant blood loss (ie, > 500 mL) within 3 months prior to the first study drug administration, and /or receipt of a blood transfusion within 1 year of first study drug administration.
25. Plasma donation within 7 days prior to the first administration of study drug.
26. Any of the following:

    1. OTC medication, herbal remedies, supplements, vitamins, or other substances from 7 days prior to first administration of study drug and during course of study without prior approval of the PI and CRO Medical monitor (with the exception of paracetamol use [maximum 2 g daily] for treatment of analgesia, ibuprofen use from Day 29, and nasal decongestant use from Day 29 [eg, phenylephrine hydrochloride, pseudoephedrine, naphazoline hydrochloride]).
    2. Unwilling to refrain from prohibited medication for study duration.
27. Use of ß-blockers within 30 days prior to first administration of study drug, or anticipated use of ß-blocker medication during the study period.
28. Anticipated use of sildenafil (Viagra®), tadalafil (Cialis®), or vardenafil (Levitra®) during the study period.
29. Anticipated using organic nitrate preparations (eg, nitroglycerin, isosorbide mononitrate, isosorbide dinitrate, pentaerythritol) during the study period.
30. Positive urine drugs screen or alcohol breath test at Screening or Day -1.
31. History of substance abuse or dependency or history of illicit drug use over the last 1 year (by self-declaration).
32. Any of the following:

    1. Regular alcohol consumption defined as > 14 standard units per week for females and > 21 standard units per week for males (where 1 standard unit = 360 mL of beer, 30 mL of 40% spirit or a 150 mL glass of wine) or > 4 standard units on any single day.
    2. Unwilling to abstain from alcohol beginning 48 hours prior to the first administration of study drug until participant check-out from the CRU.
33. Any of the following:

    1. Unwilling to abstain from caffeine (eg, coffee, tea, caffeine-containing sodas and colas) beginning 48 hours prior to the administration of the study drug and at anytime while domiciled at the CRU.
    2. Unwilling to limit the intake of caffeine beverages to < 5 cups/day from time of CRU discharge until the angiotensinogen level has returned to > 50% predose Baseline level or until at least Day 365 whichever comes first.
    3. Unwilling to abstain from xanthine-containing products (eg, chocolate) at any time while domiciled at the CRU.
34. Unwilling to refrain from strenuous exercise (including weightlifting) for 96 hours prior to each blood collection for clinical laboratory tests.
35. Employed (or is intending to be employed) as a shift worker from Screening until the angiotensinogen level has returned to > 50% predose Baseline level or until at least Day 365 whichever comes first. A shift worker is defined as a person who is employed at times falling within one of the following periods (Australian Government Fair Work Ombudsman):

    1. A night shift (commencing at or after 3 pm and before 11 pm).
    2. An early morning shift (commencing at or after 11 pm and before 4.30 am).
    3. A morning shift (commencing at or after 4.30 am and before 6.30 am).
36. Tattoos, scarring or birthmarks on the abdomen, upper arms or upper thighs that would affect the assessment of injection site reactions in the opinion of PI (or designee).
37. Anything that the PI considers that would jeopardize the safety of the participant, prevent complete participation in the study, or compromise interpretation of study data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Assess safety of ART101 by the incidence of adverse events, adverse events of special interest and SAEs | Up to Day 365 post first dose administration
Number of participants with abnormal laboratory values and/or adverse events that are related to treatment | Up to Day 365 post first dose administration
  Fasting serum chemistry, fasting hematology, fasting coagulation, fasting LFTs, fasting lipid panel, fasting glycemic assessment, urinalysis will be assessed.
Change in pharmacodynamics of ART101 by noting change from baseline of serum angiotensinogen. | Day 8, Day 15, Day 22, Day 29, Day 43, Day 57, Day 85 (~3 Months), Day 127, Day 169 (6 Months), Day 260 (9 Months) and Day 365 (12 Months) post first dose administration.

SECONDARY OUTCOMES:
PK Parameters: Maximum Concentration (Cmax) | Samples will be collected at 9 timepoints from pre-dose on Day 1, 2 timepoints on Day 2 and Day 8 post dosing
PK Parameters: Time for maximum concentration (Tmax) | Samples will be collected at 9 timepoints from pre-dose on Day 1, 2 timepoints on Day 2 and Day 8 post dosing
PK Parameters: Area under the curve (AUC) | Samples will be collected at 9 timepoints from pre-dose on Day 1, 2 timepoints on Day 2 and Day 8 post dosing
PK Parameters- Elimination half-life (t½) | Samples will be collected at 9 timepoints from pre-dose on Day 1, 2 timepoints on Day 2 and Day 8 post dosing
PK parameters: Apparent terminal elimination rate (λz ) | Samples will be collected at 9 timepoints from pre-dose on Day 1, 2 timepoints on Day 2 and Day 8 post dosing
PK parameters: Volume of distribution (Vz/F) | Samples will be collected at 9 timepoints from pre-dose on Day 1, 2 timepoints on Day 2 and Day 8 post dosing
Urine PK parameters: Renal Clearance (Ae) | Urine will be collected between 0 to 6 hours, 6 to 12 hours, 12 to 24 hours, 24 to 28 hours and Day 8 following study drug injection
Urine PK parameters: Fraction of drug excreted in urine (fe) | Urine will be collected between 0 to 6 hours, 6 to 12 hours, 12 to 24 hours, 24 to 28 hours and Day 8 following study drug injection
Urine PK parameters: Renal Clearance (CLr) | Urine will be collected between 0 to 6 hours, 6 to 12 hours, 12 to 24 hours, 24 to 28 hours and Day 8 following study drug injection

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - University of Sunshine Coast, Morayfield, Queensland
  - CMAX Clinical Research Central, Adelaide, South Australia
  - CMAX Clinical Research Fusion, Norwood, South Australia

IPD SHARING:
Plan to Share IPD: No